CLINICAL TRIAL: NCT04651686
Title: Effect of Preoperative Three-dimensional Reconstruction and Intraoperative Protection of Bronchial Artery on Cough After Thoracoscopic Pneumonectomy
Brief Title: Effect of Bronchial Artery Protection on Cough After Thoracoscopic Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20201114
Record Dates: First submitted 2020-11-22; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Cough
Keywords: Bronchial artery; Postoperative cough; three-dimensional reconstruction; Thoracoscopic surgery
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Sixty patients with thoracoscopic lobectomy and systemic lymph node dissection were selected from the same surgical group in the thoracic surgery department of the First Affiliated Hospital of Suzhou University from August 1, 2020 to October 31, 2020. According to the random number grouping method, they were divided into two groups: the bronchial artery protection group (the experimental group) and the conventional surgical treatment group (the control group). In the experimental group, 64 slice spiral CT was used for chest enhanced CT examination before operation, and mimics software was used for 3D reconstruction of bronchial artery. During the operation, the bronchial artery was protected according to the preoperative three-dimensional reconstruction image during lymph node dissection. In the control group, three-dimensional reconstruction of bronchial artery was not performed before operation, and lobectomy and systematic lymph node dissection were performed routinely
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchial artery protection (Experimental): All patients underwent chest enhanced CT examination with 64 slice spiral CT before operation. The bronchial artery was reconstructed by Mimics software. The bronchial artery was protected according to the preoperative three-dimensional reconstruction image during the lymph node dissection
  Interventions: Other: Preoperative three-dimensional reconstruction and intraoperative protection of bronchial artery

INTERVENTIONS:
Other: Preoperative three-dimensional reconstruction and intraoperative protection of bronchial artery — All patients underwent chest enhanced CT examination with 64 slice spiral CT before operation. The bronchial artery was reconstructed by Mimics software. The bronchial artery was protected according to the preoperative three-dimensional reconstruction image during the lymph node dissection

SUMMARY:
The postoperative complications of thoracoscopic radical surgery for lung cancer mainly include postoperative bleeding, pulmonary infection, chylothorax, nerve injury, pulmonary embolism, arrhythmia, postoperative cough, bronchopleural fistula and so on. Among them, postoperative cough is one of the most common complications after lung surgery, and the incidence of postoperative cough is 25% - 50%. Cough after pneumonectomy can last for a long time, which affects the rapid recovery of patients after surgery, and brings serious adverse effects to the physiological, psychological and social functions of patients.

DETAILED DESCRIPTION:
After pneumonectomy cough on patients' daily life will bring different degrees of adverse effects, so through certain methods to intervene, in order to reduce the incidence of postoperative cough, accelerate the rapid recovery of patients after surgery, improve the quality of life of patients, which should also be worthy of attention of surgeons. In recent years, the research on intervention measures and treatment methods to reduce cough after thoracoscopic lobectomy is mainly focused on drug treatment, traditional Chinese medicine treatment, surgical operation and anesthesia intervention. However, the research on reducing postoperative cough by improving surgical operation is rare. The purpose of this prospective study was to investigate whether preoperative three-dimensional reconstruction and intraoperative protection of bronchial artery can reduce the severity of cough after thoracoscopic lobectomy, so as to further explore the effective intervention measures of postoperative cough and enrich the concept of accelerated rehabilitation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no matter male or female;No cough symptoms within two weeks before operation; Lung adenocarcinoma confirmed by pathology;Operation method: thoracoscopic lobectomy + systematic lymph node dissection；Preoperative abdominal B-ultrasound, skull CT / MRI, bone scan or PET / CT to exclude distant metastasis; ECG, lung function, cardiac ultrasound evaluation can tolerate the operation

Exclusion Criteria:

* There were cough caused by respiratory diseases, pharyngitis and rhinitis before operation; Pneumonia was indicated by chest X-ray or chest CT in recent month;Thoracoscopic surgery was converted to thoracotomy;Pulmonary arteriovenous angiography could not be performed in patients with allergy to contrast medium; Patients and their families refused to be enrolled and followed up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cough | It lasted for 14 days from the first day to two weeks after operation
  Cough visual analogue scale (VAS) was used to evaluate the diagnosis of cough. Vas is a linear scoring method, using 0-100 mm scale, 0 means no cough, 100 means the most serious cough. Patients are required to mark the severity of cough on the scale line according to their own perception of cough, and measure the distance from the starting point to the marking point as a score. The higher the score is, the more serious the cough is. When the scale reaches 60mm, the patient can be diagnosed as postoperative cough.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhao, Study Director — The First Affiliated Hospital of Soochow University
Locations (1):
- Li Chang, Suzhou, Jiangsu, China

REFERENCES:
- [Background] Morita Y, Takase K, Ichikawa H, Yamada T, Sato A, Higano S, Takahashi S. Bronchial artery anatomy: preoperative 3D simulation with multidetector CT. Radiology. 2010 Jun;255(3):934-43. doi: 10.1148/radiol.10081220. PMID 20501731
- [Background] Zhang M, Liu D, Wu W, Zhang H, Mao N. Preoperative 3D-CT bronchography and angiography facilitates single-direction uniportal thoracoscopic anatomic lobectomy. Ann Transl Med. 2019 Oct;7(20):526. doi: 10.21037/atm.2019.09.135. PMID 31807508
- [Background] Anuradha C, Shyamkumar NK, Vinu M, Babu NR, Christopher DJ. Outcomes of bronchial artery embolization for life-threatening hemoptysis due to tuberculosis and post-tuberculosis sequelae. Diagn Interv Radiol. 2012 Jan-Feb;18(1):96-101. doi: 10.4261/1305-3825.DIR.3876-11.2. Epub 2011 Jun 15. PMID 21678246
- [Background] Zhu YF, Wu SB, Zhou MQ, Xie MR, Xiong R, Xu SB, Xu GW. Increased expression of TRPV1 in patients with acute or chronic cough after lung cancer surgery. Thorac Cancer. 2019 Apr;10(4):988-991. doi: 10.1111/1759-7714.13042. Epub 2019 Mar 18. PMID 30883022
- [Background] Funami Y, Okuyama K, Shimada Y, Isono K. Anatomic study of the bronchial arteries with special reference to their preservation during the radical dissection of the upper mediastinum lymph nodes. Surgery. 1996 Jan;119(1):67-75. doi: 10.1016/s0039-6060(96)80216-9. PMID 8560389